CLINICAL TRIAL: NCT07227142
Title: NOICE: A Prospective, Randomized, Crossover Study (NOICE vs. Nothing)
Brief Title: IceBath: NOICE vs Nothing
Acronym: NOICE-Icebath
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 83700
Record Dates: First submitted 2025-11-05; First posted 2025-11-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pain
Keywords: non-visual immersive technology-based audio biofeedback
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Participants first perform the task with non-visual immersive technology-based audio biofeedback using the dominant hand, followed by without non-visual immersive technology-based audio biofeedback using the non-dominant hand.
  Interventions: Behavioral: Non-visual immersive technology-based audio biofeedback intervention; Behavioral: Control (No non-visual immersive technology-based audio biofeedback)
- Group 2 (Experimental): Participants first perform the task with non-visual immersive technology-based audio biofeedback using the non-dominant hand, followed by without non-visual immersive technology-based audio biofeedback using the dominant hand.
  Interventions: Behavioral: Non-visual immersive technology-based audio biofeedback intervention; Behavioral: Control (No non-visual immersive technology-based audio biofeedback)
- Group 3 (Experimental): Participants first perform the task without non-visual immersive technology-based audio biofeedback using the dominant hand, followed by with non-visual immersive technology-based audio biofeedback using the non-dominant hand.
  Interventions: Behavioral: Non-visual immersive technology-based audio biofeedback intervention; Behavioral: Control (No non-visual immersive technology-based audio biofeedback)
- Group 4 (Experimental): Participants first perform the task without non-visual immersive technology-based audio biofeedback using the non-dominant hand, followed by with non-visual immersive technology-based audio biofeedback using the dominant hand.
  Interventions: Behavioral: Non-visual immersive technology-based audio biofeedback intervention; Behavioral: Control (No non-visual immersive technology-based audio biofeedback)

INTERVENTIONS:
Behavioral: Non-visual immersive technology-based audio biofeedback intervention — Participants receive real-time auditory feedback during cold pain endurance tasks.
Behavioral: Control (No non-visual immersive technology-based audio biofeedback) — Participants complete the same cold pain endurance tasks without any non-visual immersive technology-based auditory feedback.

SUMMARY:
This prospective, randomized, 2-period crossover study seeks to evaluate the effect of the non-visual immersive technology-based audio biofeedback intervention, delivered through devices such as NOICE device or Quest 3, on cold pain threshold within participants.

DETAILED DESCRIPTION:
This study addresses the research gap in understanding how non-visual immersive technology-based audio biofeedback intervention impacts pain perception in clinical settings. It is important to explore this because non-visual immersive technology-based audio biofeedback intervention may serve as a non-pharmaceutical, non-visual immersive technology-based audio biofeedback alternative to traditional visual-based distraction methods like virtual reality.

The investigators hypothesize that participants using the non-visual immersive technology-based audio biofeedback device will report an increased pain threshold compared to not using the device. This knowledge could improve information on the perception of pain for participant who prefer not to use Virtual Reality (VR) headsets.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and older
* English-speaking
* Intact hearing
* No self-reported or clinically diagnosed acute or chronic medical conditions that may affect safe participation

Exclusion Criteria:

* Use chronotropic heart medications
* Use pain medications
* Current hearing loss
* Currently taking beta blockers, or opioids or other prescription pain medications
* History of chronic pain or acute pain syndromes

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | Immediately after intervention
  Pain sensitivity will be measured by Numerical Rating Pain Scale. Participants will rank pain scores on a sliding scale from 0 = No Pain to 10 = Worst possible pain

SECONDARY OUTCOMES:
Anxiety Level | Immediately after intervention
  Participants will complete the Visual Analog Scale for Measuring Anxiety (VAS-A) immediately following each group of levels tests, where they will rank anxiety scores on a sliding scale from 0 = No anxiety/fear to 100 = Worst possible anxiety/fear
Cold pain endurance | Periprocedural
  To evaluate Cold Pain Endurance, total time (in seconds) that the participant's hand remains immersed in ice water will be recorded. Start time is defined as the moment immediately prior to immersion, and stop time as the moment the hand is withdrawn.
ISO Ergonomic scale | immediately after intervention
  The scale has 6 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
System Usability Scale (SUS) Score | immediately after intervention
  The scale has 10 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
Device satisfaction | immediately after intervention
  To evaluate the overall impact of device satisfaction of the spatial audio stimulation device, participants will complete the Patient Technology Satisfaction Survey. Participants will rank each factor on a Likert scale from 1 = not at all to 5 = completely.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Childrens Hospital Stanford, Palo Alto, California, United States